CLINICAL TRIAL: NCT03030820
Title: Oral Gut Liver Axis in Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HM20006081
Record Dates: First submitted 2017-01-05; First posted 2017-01-25 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Cirrhosis; Periodontitis; Gingivitis
Keywords: cirrhosis; Periodontitis; oral health; gingivitis; inflammation
MeSH Terms: conditions — Fibrosis; Periodontitis; Gingivitis; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dental cleaning (Experimental): Patients with cirrhosis and healthy controls will undergo dental examination and subsequent dental cleaning if necessary.
  Interventions: Procedure: Dental Cleaning

INTERVENTIONS:
Procedure: Dental Cleaning — This is standard of care dental cleaning as is guided by the initial dental evaluation

SUMMARY:
This will be a prospective study of cirrhotics and healthy controls comparing their oral microbiota, endotoxemia and systemic inflammation at baseline and at 30 days after clinically indicated systematic oral cleansing and interventions as well as 3-month hospitalizations post-cleaning.

DETAILED DESCRIPTION:
This will be a prospective study of cirrhotics and healthy controls comparing their oral microbiota, endotoxemia and systemic inflammation at baseline and at 10 and 30 days after clinically indicated systematic oral cleansing and interventions as well as 3-month hospitalizations post-cleaning.

The investigators will recruit cirrhotic subjects and age- matched healthy controls from the hepatology clinics. Subjects will be informed regarding the study and will give the investigators a written informed consent.

After informed consent and evaluation of eligibility, subjects will be asked to complete an oral health questionnaire and sample collection during the recruitment visit. Patients will then be scheduled for a dental exam during a separate screening visit up to 7 days after this recruitment visit at the Dental Clinics.

At this time patients will undergo cognitive testing consisting of a validated cognitive battery of PHES (psychometric hepatic encephalopathy score) and EncephalApp stroop. In addition, they will undergo Sickness Impact Profile (a quality of life questionnaire).

During dental exam which will be done during screening visit, the subject will undergo comprehensive oral evaluation which will include dental xrays (as needed) which are part of the study, periodontal examination (determination of pocket depth, clinical attachment levels, bleeding on probing, plaque index) and recording of caries and oral soft tissue lesions. Dental cleaning is part of the study protocol and not intended to fully treat the patient's periodontal and dental diseases. Therefore no follow-up dental visits will be scheduled in the dental clinics after completion of dental cleansing.

The patients who do not qualify for the study will be informed of the findings by the dental professionals and subsequently the patients need to make arrangements for their dental treatment needs.

The study will include cirrhotic patients with/without hepatic encephalopathy. Subjects will then be scheduled for dental cleaning which could occur over 1 or 2 visits as determined during the screening exam.

Before the initiation of oral therapy, plaque and gingival crevicular samples will be collected for microbiota. The subjects will receive deep dental cleanings (scaling and root planing) and oral hygiene instructions as per clinical indication.

Subjects will then be followed at day 10 for clinical exam and day 30 at which point stool, saliva and blood samples for the similar analyses as before will be collected. There will be no more dental examinations after the initial assessment and treatment. We will repeat the cognitive testing at day 30 using alternate forms of the same cognitive tests and also repeat quality of life testing at day 30 .

The investigators will also follow them for up to 3 months post-cleaning for hospitalizations using active chart review and follow-up

ELIGIBILITY:
Inclusion criteria:

Cirrhotic subjects:

1. Age 21-75 years
2. Able to give informed consent
3. Cirrhosis diagnosed using biopsy or suggestive radiological features or endoscopic evidence of varices in a subject with chronic liver disease

Healthy controls:

1. Age 21-75 years
2. Able to give informed consent
3. Without chronic diseases

Exclusion Criteria:

Exclusions for all subjects (will be done at the screening visit at both clinics)

1. Current use of absorbable antibiotics (use of antibiotics within 4 weeks)
2. Diagnosed with severe chronic or aggressive forms of periodontitis based on American Academy of Periodontology Classification (5)
3. Presence of more than 2 severe cavitated caries lesions
4. Presence of oral soft-tissue lesions such as ulcers
5. Presence of abscesses
6. Unclear diagnosis of cirrhosis (for cirrhotics)
7. Edentulous or less than 20 natural teeth
8. Smoking, oral tobacco and alcohol abuse within 3 months
9. Prisoners
10. Pregnant women
11. INR(international normalized ratio) >1.5
12. Platelet count <50,000
13. Diagnosed bleeding disorders
14. Patients on anti-coagulation
15. Patients who will otherwise be eligible for prophylactic antibiotics before dental cleaning
16. Last dental cleaning within 3 months of study.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-10; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change in serum endotoxin | 30 days
  Relative change in serum endotoxin levels using LAL (limulus amebocyte lysate) assay will be measured before/after cleaning and between groups

SECONDARY OUTCOMES:
Change in performance on two batteries of Cognitive function | 30 days
  Relative change in PHES battery (total standard deviations above normal performance)and EncephalApp Stroop values (seconds taken) will be measured before/after cleaning and between groups
Change in systemic inflammatory cytokines in the blood | 30 days
  Relative change in pg/ml of serum IL-6 (interleukin), IL-1b (interleukin) using ELISA assays will be measured before/after cleaning and between groups
All-cause Hospitalizations | 3 months
  All-cause, liver-related and elective hospitalizations at 3 months will be studied and compared between groups
Change in microbiota composition in the saliva and stool | 30 days
  Relative change in microbial composition using 16SrRNA multi-tagged sequencing in stool and saliva will be measured before/after cleaning and between groups
MELD (model for end-stage liver disease) score change in the cirrhosis group | 30 days
  Relative change in MELD score will be analyzed in cirrhotic patients before/after cleaning
Quality of life changes | 30 days
  Changes in quality of life using Sickness Impact Profile will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Jasmohan Bajaj, MD, Principal Investigator — VCU medical Center
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No